CLINICAL TRIAL: NCT01409473
Title: A Prospective Protocol of Stereotactic Body Irradiation With Concurrent Intraprostatic Lesion Boost Utilizing Intensity Modulated Radiotherapy for Patients With Low- and Intermediate-Risk Prostate Cancer
Brief Title: Stereotactic Body Radiotherapy (SBRT) With Concurrent Boost for Low- and Intermediate-Risk Prostate Cancer
Acronym: Prostate SBRT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Rocky Mountain Cancer Centers (Other)
Collaborators: Dr. Dennis Carter (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 511-03; WIRB #20111125 (Other: Western IRB)
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Stereotactic body radiotherapy; Radiosurgery; Intensity-modulated radiotherapy; SBRT; IMRT; Early-stage prostate cancer; Low-risk prostate cancer; Intermediate-risk prostate cancer; Intraprostatic lesions; IPL
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostate SBRT (Experimental): Prostate SBRT with concurrent boost to intraprostatic lesion (IPL) will be delivered in 5 fractions using intensity-modulated radiotherapy planning techniques.
  Interventions: Radiation: Prostate SBRT with concurrent boost to intraprostatic lesion(s)

INTERVENTIONS:
Radiation: Prostate SBRT with concurrent boost to intraprostatic lesion(s) — 40 Gy in 5 fractions to prostate for low-risk and 45 Gy in 5 fractions to prostate for intermediate-risk patients, and 50 Gy in 5 fractions to intraprostatic lesion(s), delivered over 10-14 days on preferably every other day.
  Other Names: Stereotactic surgery to the prostate

SUMMARY:
The purpose of this study is to determine whether stereotactic body radiation therapy (SBRT) with simultaneous boost (higher radiation dose) to areas within the prostate with more prominent cancerous growth (intraprostatic lesions) utilizing intensity modulated radiotherapy (IMRT) planning techniques is a safe and effective treatment in patients with low- and intermediate-risk localized prostate cancer.

DETAILED DESCRIPTION:
Standard external beam radiation therapy (EBRT) for low- to intermediate-risk prostate cancer involves several weeks of daily treatment sessions. Stereotactic body radiation therapy (SBRT) is a newer form of EBRT that gives fewer treatments but higher doses of radiation per treatment. In many patients there are certain areas within the prostate with more prominent cancerous growth (intraprostatic lesions), which may require higher doses of radiation (boost) to treat effectively. This study will treat the prostate with simultaneous boost(s) to intraprostatic lesion(s) in 5 treatments over 10-14 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of prostate adenocarcinoma within one year
* Gleason Score 2-7
* Clinical T-stage T1b-T2c (AJCC 7th Edition)
* Clinical Nx or N0, and Mx or M0
* PSA < 20 ng/mL
* Low or intermediate risk according to NCCN guidelines: Low: Clinical Stage (CS) T1b-T2a and Gleason 2-6 and PSA < 10 ng/ml; Intermediate: CS T2b-T2c and Gleason 2-6 and PSA < 10 ng/ml, or CS T1b-T2a and Gleason 7 and PSA < 10 ng/ml, or CS T1b-T2a and Gleason 2-6 and PSA 10-20ng/mL
* ECOG performance status 0 or 1
* Has had a pre-treatment PSA drawn within a month of the beginning of protocol therapy
* If androgen-deprivation therapy (ADT) has been initiated, must have a documented pre-ADT PSA; this baseline PSA should not be obtained during following periods: 1) 10-day period following prostate biopsy; 2) within 30 days after discontinuation of finasteride; or 3) within 90 days after discontinuation of dutasteride.
* Has completed a baseline health-related quality of life assessment Extended Prostate Cancer Index Composite questionnaire (EPIC-26)
* Has had a history and physical examination (including digital rectal examination and a formal morbidity assessment via the ACE-27) within 60 days
* Morbidity score (via the ACE-27) of none (0), mild (1) or moderate (2)
* Willing and able to use adequate contraception during protocol treatment and for 3 months after the completion of protocol treatment

Exclusion Criteria:

* Invasive (carcinoma in situ is allowed) solid or hematologic malignancy (other than this prostate cancer, or basal or squamous skin cancers) in the last 5 years
* Prior prostatectomy or cryotherapy of the prostate
* Prior radiotherapy to the prostate or lower pelvis
* Prior or concurrent cytotoxic chemotherapy for prostate cancer (prior chemotherapy for a different cancer is allowed)
* Implanted hardware near the planning target volume that would prohibit appropriate treatment planning or treatment delivery in the investigator's opinion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2018-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Biochemical disease-free survival | 5-8 years
  Biochemical Disease-Free Survival (bDFS), the time from completion of protocol treatment to the documented PSA rise of 2 ng/mL above the PSA nadir reached after treatment.

SECONDARY OUTCOMES:
Grade 2 or higher acute gastrointestinal, genitourinary, and erectile toxicities | 30 days from completion of protocol radiotherapy
  Grade 2 or higher acute gastrointestinal, genitourinary, and erectile toxicities, graded per CTCAE 3.0. Acute adverse events will be recorded as the first occurrence of worst severity of the adverse event ≤ 30 days from completion of protocol radiotherapy.
Grade 3 or higher late gastrointestinal, genitourinary, and erectile toxicities | >30 days to 5 years from completion of protocol radiotherapy
  Grade 3 or higher late gastrointestinal, genitourinary, and erectile toxicities, graded per CTCAE 3.0. Late adverse events are defined as the first occurrence of a late grade 3+ adverse event > 30 days from completion of protocol radiotherapy.
Freedom from failure | 5-8 years
  Freedom from failure, defined as the time from the first date of radiation to first event of biochemical failure (nadir + 2 ng/mL), local recurrence, regional recurrence, or distant disease as defined below.
Local recurrence-free survival | 5-8 years
  Local recurrence-free survival, defined as the time from the first date of radiation to first pathologic confirmation of in-prostate tumor recurrence. The local recurrence will be dated when the palpable progression was first identified. In the event of biochemical failure followed by negative metastatic workup and positive biopsy for in-prostate recurrence, the local recurrence will be dated the date of the documented biochemical failure.
Distant disease-free survival | 5-8 years
  Distant disease-free survival, defined as the time from the first date of radiation to first documentation of metastatic disease by any method, regardless of the occurrence of any intervening local or regional failure or non-prostate second primary cancer. If metastatic diagnosis was prompted by biochemical failure, distant recurrence will be dated the date of biochemical failure.
Cause-specific survival | 5-8 years
  A death will be deemed a prostate cancer specific death if death is due to prostate cancer or a complication from treatment.
Overall survival | 8-10 years
  Overall survival, defined as the time from the first date of radiation to death due to any cause.
Health-related quality of life | 2-3 years
  Health-related quality of life (HRQOL), measured with the Extended Prostate Cancer Index Composite questionnaire - short form (EPIC-26).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Leonard, MD, Principal Investigator — Rocky Mountain Cancer Centers
Locations (2):
- United States (2):
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Littleton, Littleton, Colorado